CLINICAL TRIAL: NCT06703424
Title: Investigating the Acute Effects of Light Intensity Physical Activities on Pre-frontal Cortical Activation, Cognitive Function, Sleepiness and Back Pain Among Physically Inactive University Students
Brief Title: Effects of Light Intensity Physical Activities on Pre-frontal Cortical Activation, Cognitive Function, Sleepiness and Back Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chia Yong Hwa Michael (Other)
Collaborators: Sendai University (Unknown)
Responsible Party: Sponsor-Investigator, Chia Yong Hwa Michael, Principal Investigator, Nanyang Technological University
Organization: Nanyang Technological University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: NanyangTU
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Pre-frontal Cortical Oxygenated and Deoxygenated Hemoglobin Levels
Keywords: light-intensity exercise; pre-frontal cortical activation; executive functioning; university students; inactive
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Two-arm intervention, crossover study design
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sit-cycling (Experimental): Sit-cycling on a seat-cycle for 5 mins
  Interventions: Other: Sit-cycling
- Stand-twisting (Experimental): Stand-twisting on a stand-twister for 5 mins
  Interventions: Other: Stand-twisting
- Sitting only (No Intervention): Sitting only for 5 mins

INTERVENTIONS:
Other: Sit-cycling — Sit-cycling for 5 mins
  Arms: Sit-cycling
Other: Stand-twisting — Stand-twisting for 5 mins
  Arms: Stand-twisting

SUMMARY:
The objective of this randomised controlled trial is to examine the acute effects of two novel light intensity exercise (sit-cycling and stand-twisting) on prefrontal cortical blood oxygenation, executive functioning, sleepiness and back pain among inactive university students.

The main questions it aims to answer are:

* What are the changes in oxygenated haemoglobin (O2Hb) and deoxygenated hemoglobin (HHb) levels in the prefrontal cortex from baseline to immediately after and 20 minutes after a 5-min bout of S-C and S-T compared to sitting for the same duration?
* What are the changes in executive functioning, specifically, n-back test and Word Colour Stroop test performance from baseline to immediately after and 20 minutes after a bout of S-C and S-T compared to sitting for the same duration?
* How does participants' self-rated daytime sleepiness and back pain after a bout of S-C and S-T compare to sitting for the same duration?

Participants will:

* Perform sit-cycling or stand-twisting for 5 mins (experimental condition) and sit for 5 mins (control condition)
* Wear the functional near-infrared spectroscopy cap on their head throughout the measurements
* Complete 1-back, 2-back test and Word Colour Stroop before, immediately after and 20 minutes after experimental/ control condition
* Have their blood pressure, heart rate taken by a smartwatch
* Complete a daytime sleepiness questionnaire and a back pain questionnaire

ELIGIBILITY:
Inclusion Criteria:

* NTU-NIE university student, between 21 and 30 years old, do not meet physical activity guidelines (150 mins of weekly MVPA)

Exclusion Criteria:

* taking blood-pressure lowering medication
* physically active (150 mins or more of weekly MVPA)
* deemed not physically fit to participate in physical activity based on responses to Get Active Questionnaire

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2024-08-11 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
1-back test accuracy (%) | Pretest, post-test 1 (immediately after experimental condition) and post-test 2 (after post-test 1)
  Number of correct trials (correct recall)
1-back test reaction time (ms) | Pretest, post-test 1 (immediately after experimental condition) and post-test 2 (after post-test 1)
  Average reaction time across trials
2-back test accuracy (%) | Pretest, post-test 1 (immediately after experimental condition) and post-test 2 (after post-test 1)
  Number of correct trials (correct recall)
2-back test reaction time (ms) | Pretest, post-test 1 (immediately after experimental condition) and post-test 2 (after post-test 1)
  Average reaction time across trials
Colour Word Stroop test accuracy (congruent) (%) | Pretest, post-test 1 (immediately after experimental condition) and post-test 2 (after post-test 1)
  Number of correct trials recall
Colour Word Stroop test accuracy (incongruent) (%) | Pretest, post-test 1 (immediately after experimental condition) and post-test 2 (after post-test 1)
  Number of correct trials recall
Colour Word Stroop test reaction time (congruent) (ms) | Pretest, post-test 1 (immediately after experimental condition) and post-test 2 (after post-test 1)
  Average reaction time across trials
Colour Word Stroop test reaction time (incongruent) (ms) | Pretest, post-test 1 (immediately after experimental condition) and post-test 2 (after post-test 1)
  Average reaction time across trials
pre-frontal cortical oxygenated hemoglobin levels (micrometre) | Pretest, post-test 1 (immediately after experimental condition) and post-test 2 (after post-test 1)
  measured by functional near infrared spectroscopy
pre-frontal cortical deoxygenated hemoglobin levels (micrometre) | Pretest, post-test 1 (immediately after experimental condition) and post-test 2 (after post-test 1)
  measured by functional near infrared spectroscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Block 5 Physical Education and Sport Science, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Individual participant data constitute as personal data. Under the Singapore Personal Data Protection Act, it is mandatory that individually identifiable data are to be kept confidential.